CLINICAL TRIAL: NCT00059020
Title: EGF Polymorphisms and Gliomagenesis
Brief Title: The Role of Gene Changes in Brain Tumor Formation and Growth
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030160; 03-N-0160
Record Dates: First submitted 2003-04-16; First posted 2003-04-16 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2004-11

CONDITIONS: Glioma
Keywords: Glioma; Brain Tumor; Epidermal Growth Factor; Polymorphisms
MeSH Terms: conditions — Glioma; Brain Neoplasms

SUMMARY:
This study will examine tissue from gliomas (a type of brain tumor) removed during surgery for gene mutations, or changes, thought to be involved in tumor formation and growth. One common gene mutation causes the receptor for a protein called epidermal growth factor (EGF) to be in an active state all of the time, allowing uncontrolled cell growth that can lead to tumor formation. This study will analyze blood and tumor tissue samples from patients with gliomas for:

* Changes in the EGF gene in the tumor
* Changes in other genes, such as that for the EGF receptor (EGFR)
* Changes in levels of EGF and EGFR, and in other proteins and genes that respond to changes in the levels of these proteins in the tumor
* Changes in the EGF gene and protein in the blood

The study will also determine if production of EGF and EGFR obtained from glioma and from blood cells derived from the tumor can be altered in the laboratory to grow indefinitely in culture.

Patients between 18 and 75 years of age with a brain tumor that requires surgical treatment may be eligible for this study.

Participants will be admitted to the NIH Clinical Center for about 3 to 10 days. They will have a physical and neurological examination, blood and urine tests, other tests, if medically necessary, and will be evaluated and prepared for surgery. During surgery, as much of the tumor as possible will be removed. A small amount of the tumor tissue will be collected for this study. No tissue will be removed for this study that would not otherwise have been removed. Some of the tissue will be used to culture glioma cells and the rest will be frozen and stored for examination, as described above. If any normal-appearing brain tissue is removed during surgery in order to enhance safety in removing the tumor, the normal tissue will be studied as well. Brain tissue that appears normal will not be removed strictly for research.

During surgery and the day after surgery, a blood sample will be drawn from a catheter (plastic tube) that was placed in an artery or vein for surgery. If catheters are no longer in place, blood will be drawn through a needle in a vein.

DETAILED DESCRIPTION:
The epidermal growth factor (EGF) is an important biological mediator of normal growth and repair and is critical to epithelial tissue development and maturation of the central nervous system, among other functions. EGF is a natural focus of interest in cancer research because of its influence over mitogenesis, proliferation, and tumorigenesis. In addition, unregulated expression of its receptor, EGFR, has been identified as a common event in neoplastic transformation. In patients with the most malignant primary tumor of the brain, the glioblastoma multiforme (GBM), alterations in the EGFR or in its expression levels have been identified in approximately 50% of patients. We postulate that EGF-EGFR interactions may be important for the development, progression, and prognosis of human gliomas and that alterations of the EGF gene may predict the potential for glioma progression and the severity of disease.

Patients suspected of having, or with prior biopsy proof of, a WHO grade II-IV central nervous system (CNS) glial tumor(s) seen in the Surgical Neurology Branch, NINDS, will be considered for entry into this study. Tissue samples of tumor resected as part of standard care will be collected at surgery and preserved for research. Blood samples will also be collected. Blood will also be collected from anonymous normal volunteers who donate blood at the NIH Blood Bank; these anonymous donors will serve as controls.

ELIGIBILITY:
INCLUSION CRITERIA:

Radiographic evidence of a primary glial neoplasm of the CNS (WHO grade II-IV) or any patient with known primary neoplasms of the CNS.

Medically indicated diagnostic and/or therapeutic tumor resection.

Informed consent from patient, age 18 or older to 75 years of age.

Females of child-bearing capacity: Pregnant women will be entered into the study for tumor collection, but blood will not be drawn at the time of surgery. Six weeks or more after the completion of pregnancy, these women will be contacted and 10cc (2 tsp) of blood will be collected for genotyping.

No racial or ethnic group or gender is excluded.

EXCLUSION CRITERIA:

Inability to provide informed consent prior to surgery.

Medical conditions that cannot be corrected prior to surgery that would be standard contraindications for neurosurgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 344
Dates: Start 2003-04; Study Completion 2004-11

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Burdick JS, Chung E, Tanner G, Sun M, Paciga JE, Cheng JQ, Washington K, Goldenring JR, Coffey RJ. Treatment of Menetrier's disease with a monoclonal antibody against the epidermal growth factor receptor. N Engl J Med. 2000 Dec 7;343(23):1697-701. doi: 10.1056/NEJM200012073432305. No abstract available. PMID 11106719
- [Background] Groenen LC, Nice EC, Burgess AW. Structure-function relationships for the EGF/TGF-alpha family of mitogens. Growth Factors. 1994;11(4):235-57. doi: 10.3109/08977199409010997. PMID 7779404
- [Background] Laurence DJ, Gusterson BA. The epidermal growth factor. A review of structural and functional relationships in the normal organism and in cancer cells. Tumour Biol. 1990;11(5):229-61. PMID 2203137